CLINICAL TRIAL: NCT00873730
Title: A 12-week Randomized, Double-blind, Multicenter Pilot Study to Evaluate the Effect of Etanercept 100 mg and 50 mg Weekly in Subjects With Ankylosing Spondylitis
Brief Title: Study Evaluating Etanercept in Subjects With Ankylosing Spondylitis in Spain
Acronym: Loadet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-406
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Effect of etanercept in subjects with ankylosing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: etanercept
- 2 (Active Comparator)
  Interventions: Drug: etanercept/placebo

INTERVENTIONS:
Drug: etanercept — Etanercept 50 mg twice a week (BIW) for 12 weeks
  Arms: 1
Drug: etanercept/placebo — Etanercept 50 mg once a week (QW) and placebo once a week for 12 weeks
  Arms: 2

SUMMARY:
The purpose of this study was to evaluate efficacy and safety of etanercept 100 mg (50 mg twice a week) compared with 50 mg once a week in adult subjects with ankylosing spondylitis (AS) and previous failure to usual practice therapies in Spain.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of ankylosing spondylitis, as defined by Modified New York Criteria for Ankylosing Spondylitis.
2. Maintained inflammatory activity for more than 12 weeks defined by:·Axial forms: BASDAI higher than or equal to 4 (0-10) and at least one of the following parameters:. Global assessment of the disease by the patient higher than or equal to 4 (On a scale 0-10). Spinal pain higher than or equal to 4 on a visual analogue scale (VAS). Increase in erythrocyte sedimentation rate (ESR) and/or CRP above the normality parameters established by the laboratory.·Peripheral forms: Arthritis or enthesitis higher than or equal to 1 site and at least one of the following:. Global assessment of the disease by the patient higher than or equal to 4 (on a scale 0-10). Increase in erythrocyte sedimentation rate (ESR) and/or CRP above the normality parameters established by the laboratory
3. Failure to treatment: Failure to at least 2 NSAIDs at maximum recommended dose during at least 3 months (or a shorter time in case of intolerance, toxicity or contraindication).·In cases of ankylosing spondylitis with peripheral joint involvement, salazopyrine should have been used at a dose of 2-3 g per day and/or methotrexate (15 mg/week) for 4 months (or a shorter time in case of intolerance, toxicity or contraindication). In case of oligoarticular or localized involvement in enthesis: lack of response, at the discretion of the investigator, to local infiltrations and/or synoviorthesis.
4. Be between 18-70 years of age
5. Negative result of a pregnancy test in serum in screening visit and in urine in baseline visit, done in all women, except those surgically sterilized and those who have at least one year of menopause.
6. Sexually active women of childbearing potential must use medically acceptable contraceptive methods, including oral, injectable or implantable contraceptive methods, intrauterine devices or properly used barrier contraception. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant. This includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives.
7. Men who are not surgically sterile should agree to use reliable contraceptive methods during the study.
8. Ability to reconstitute the drug and self-inject it or have a person who can do so.
9. Capability to understand and voluntarily give written informed consent that is signed and dated, before any specific procedure of the protocol is performed.
10. Ability to store injectable test article at 2º to 8º C.

Exclusion criteria:

1. Contraindications for treatment with anti-TNF
2. Complete ankylosis of spine
3. Onset of treatment with DMARDs in the 4 weeks prior to baseline (SSZ, MTX and HCQ are permitted if the administrated dose has been maintained stable in the 4 weeks prior to baseline). Furthermore, patients with a dose of prednisone >10 mg/d or equivalent or modified in the 2 weeks prior to the baseline visit, those in whose infiltration has been performed with intraarticular corticosteroids has been performed in the 4 weeks prior to the screening visit and those who follow treatment with more than one NSAID in the 2 weeks prior to the baseline visit are excluded.
4. Previous treatment with other TNF inhibitors and other biological drugs
5. Abnormalities in hematology profiles defined by:

   * leukocytes lower than or equal to 3.5 x 10 exponent 9 /L
   * hemoglobin lower than or equal to 8.5 g/L or 5.3 mmol/L
   * hematocrit lower than or equal to 27%
   * platelets lower than or equal to 125 x 10 exponent 9 /L
   * serum creatinine higher than or equal to 175 mmol/L
   * aspartate aminotransferase and alanine aminotransferase higher than or equal to 2 times the upper limit of normality
6. Important concomitant medical conditions, such as:-Class III or IV congestive heart failure according to New York Heart Association classification-Uncontrolled arterial hypertension (defined as screening systolic blood pressure > 160 mm Hg or screening diastolic blood pressure > 100 mm Hg)-Myocardial infarction within 12 months of the screening visit or unstable angina-Severe pulmonary disease requiring hospitalization or oxygen therapy-Diagnosis of multiple sclerosis or other central nervous system demyelinating disease -Presence or history of confirmed blood dyscrasias-Cancer or history of cancer (other than resected cutaneous basal cell or squamous cell carcinoma)-Serious infection (infection requiring hospitalization and/or intravenous antibiotics) within 1 month of administration of test article administration or active infection at screening or history of recurrent or chronic infection-Open cutaneous ulcers-Patients with known chronic infections as positivity to HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) -Active tuberculosis infection (local guidelines for appropriate screening and treatment of tuberculosis in the setting of anti-TNF therapy must be followed)- Any condition that, in the investigator's judgment, might cause this study to be detrimental to the subject
7. Pregnant or breast-feeding women
8. Past or current psychiatric illness that would interfere with the subject's ability to comply with protocol requirements or give informed consent.
9. Treatment with any live (attenuated) vaccine within 4 weeks prior to baseline.
10. History of alcohol or drug abuse that would interfere with the subject's ability to comply with protocol requirements.
11. Treatment with any investigational drug within 3 months of screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Navarro-Sarabia F, Fernandez-Sueiro JL, Torre-Alonso JC, Gratacos J, Queiro R, Gonzalez C, Loza E, Linares L, Zarco P, Juanola X, Roman-Ivorra J, Martin-Mola E, Sanmarti R, Mulero J, Diaz G, Armendariz Y, Collantes E. High-dose etanercept in ankylosing spondylitis: results of a 12-week randomized, double blind, controlled multicentre study (LOADET study). Rheumatology (Oxford). 2011 Oct;50(10):1828-37. doi: 10.1093/rheumatology/ker083. Epub 2011 Jun 23. PMID 21700683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Spain from December 2006 to February 2008.
Pre-assignment Details: Patients were screened up to 6 weeks.
Groups:
- Etanercept BIW: etanercept 50 mg twice a week (BIW) for 12 weeks
- Etanercept QW: etanercept 50 mg once a week (QW) and placebo once a week for 12 weeks
Period: Overall Study
Arm/Group | Etanercept BIW | Etanercept QW
Started | 54 | 54
Completed | 48 | 49
Not Completed | 6 | 5
Not completed — Protocol Deviation | 5 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Sponsor decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept BIW | Etanercept QW | Total
Number analyzed (Participants) | 54 | 54 | 108
Age Continuous [Mean (Standard Deviation); unit: years] | 40.22 (10.36) | 42.63 (10.66) | 41.43 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Assessment in Ankylosing Spondylitis (ASAS) 20.
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients. ASAS = 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement (vs. baseline) and an absolute change ≥ 10 units on a 0-100 scale (0=no disease activity; 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
patients | 34 | 37
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.6031, Chi-squared

2. Secondary Outcome: Number of Patients Achieving Assessment in Ankylosing Spondylitis (ASAS) 40.
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients. ASAS = 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40% improvement (vs. baseline) and an absolute change ≥ 20 units on a 0-100 scale (0=no disease activity, 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
patients | 25 | 25
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.9166, Chi-squared

3. Secondary Outcome: Number of Patients Achieving Assessment in Ankylosing Spondylitis (ASAS) 50.
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients. ASAS = 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 50 = 50% improvement (vs. baseline) and an absolute change ≥ 20 units on a 0-100 scale (0=no disease activity, 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
patients | 22 | 24
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.7564, Chi-squared

4. Secondary Outcome: Number of Patients Achieving Assessment in Ankylosing Spondylitis (ASAS) 70.
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients. ASAS = 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 70 = 70% improvement (vs. baseline) and an absolute change ≥ 20 units on a 0-100 scale (0=no disease activity, 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
patients | 15 | 20
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.3266, Chi-squared

5. Secondary Outcome: Number of Patients Achieving Assessment in Ankylosing Spondylitis (ASAS) 5/6.
Description: ASAS 5/6 consists of 6 domains: the 4 used in ASAS 20 (patient global assessment of disease activity, pain, function, inflammation measured on a 0-100 scale, where 0=no disease activity, 100=high disease activity) plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). Achieving ASAS 5/6 requires a 20% improvement compared to baseline in ≥ 5 domains and no worsening in the remaining domain.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
patients | 20 | 22
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.7481, Chi-squared

6. Secondary Outcome: Number of Patients Achieving Partial Remission.
Description: Partial remission defined as a score of less than 20 units (on a scale of 0-100, where 0=no disease activity, 100=high disease activity) in each of the 4 Assessment in Ankylosing Spondylitis (ASAS) domains: patient global assessment of disease activity, pain, function, and inflammation. For scale, 100=high disease activity.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
patients | 14 | 13
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.7721, Chi-squared

7. Secondary Outcome: Change in Nocturnal Back and Overall Spinal Pain From Baseline to Week 12.
Description: Nocturnal back and overall spinal pain assessed by patients using a Visual Analog Scale (VAS) of 0 - 10 (0 = no pain and 10 = most severe pain).
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
units on scale
  Nocturnal Back Pain | -3.96 (3.15) | -4.15 (2.76)
  Overall Spinal Pain | -3.89 (2.99) | -3.53 (2.85)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Nocturnal Back Pain; Test type: Superiority or Other; p = 0.6660, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Overall Spinal Pain; Test type: Superiority or Other; p = 0.5364, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Physician and Patient Global Assessment (PGA) of Pain From Baseline to Week 12.
Description: Patient pain assessed by physician and patient using a Visual Analog Scale (VAS) of 0 - 10 (0 = none and 10 = severe).
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
units on scale
  Physician Global Assessment | -4.15 (1.77) | -4.12 (1.39)
  Patient Global Assessment | -3.67 (3.13) | -4.17 (2.69)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for the Physician Global Assessment; Test type: Superiority or Other; p = 0.9426, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for the Patient Global Assessment; Test type: Superiority or Other; p = 0.4969, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Bath Ankylosing Spondylitis Functional Index (BASFI) From Baseline to Week 12.
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in AS patients. Utilizing a VAS of 0-10 (0=easy, 10=impossible), patients answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions.
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
units on scale | -2.61 (2.64) | -2.45 (2.12)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.6687, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) From Baseline to Week 12.
Description: BASDAI is a validated self assessment tool used to determine disease activity in patients with Ankylosing Spondylitis (AS). Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) patient's answered 6 questions measuring discomfort, pain and fatigue. The BASDAI final mean score was calculated taking all 6 VAS assessments.
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 48 | 49
units on scale | -3.67 (2.18) | -3.59 (2.46)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.6739, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Bath Ankylosing Spondylitis Metrology Index (BASMI) From Baseline to Week 12.
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10.
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 46 | 45
units on scale | -0.46 (0.98) | -0.80 (1.27)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.2772, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Erythrocyte Sedimentation Rate (ESR) From Baseline to Week 12.
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube and is measured in mm/hour. Normal range is 0-30mm/h. A higher rate is consistent with inflammation.
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 47 | 46
mm/hour | -11.8 (14.47) | -16.2 (16.06)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.1560, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Ankylosing Spondylitis Quality of Life (EuroQoL) Questionnaire
Description: EuroQol questionnaire is intended to measure the quality of life by means of questions about mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Answers to every question were grouped in two main categories: with problems (having some problems or absolutely unable) or without problems.
Time Frame: 12 weeks
Population: The analysis population was the intent to treat population.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 47 | 49
patients
  Mobility Without Problems | 37 | 33
  Mobility With Problems | 10 | 16
  Self-care Without Problems | 29 | 29
  Self-care With Problems | 18 | 20
  Usual activities Without Problems | 20 | 17
  Usual activities With Problems | 27 | 32
  Pain/Discomfort Without Problems | 5 | 13
  Pain/Discomfort With Problems | 42 | 36
  Anxiety/Depression Without Problems | 28 | 32
  Anxiety/Depression With Problems | 19 | 17
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Mobility; Test type: Superiority or Other; p = 0.2099, Chi-squared
Statistical Analysis 2: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Self-care; Test type: Superiority or Other; p = 0.8009, Chi-squared
Statistical Analysis 3: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Usual activities; Test type: Superiority or Other; p = 0.4290, Chi-squared
Statistical Analysis 4: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Pain/Discomfort; Test type: Superiority or Other; p = 0.0461, Chi-squared
Statistical Analysis 5: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Anxiety/Depression; Test type: Superiority or Other; p = 0.5620, Chi-squared

14. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline to Week 12.
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline and 12 weeks
Population: The analysis population was the intent to treat population. Two scored areas had a different "Number of Participants Analyzed" in the etanercept arm. Bodily pain had 45 and Emotional role limitations had 46.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 47 | 49
units on scale
  Physical functioning | 15.53 (27.73) | 19.90 (20.73)
  Physical role limitations | 30.32 (50.79) | 32.14 (42.08)
  Bodily pain | -1.39 (22.31) | -1.43 (24.02)
  General health | 7.23 (13.22) | 9.59 (12.11)
  Vitality | 8.65 (13.61) | 12.14 (14.58)
  Social functioning | 8.24 (16.75) | 6.12 (20.59)
  Emotional role limitations | 17.39 (42.01) | 17.01 (40.89)
  Mental health | 7.34 (11.53) | 6.27 (11.02)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Physical functioning; Test type: Superiority or Other; p = 0.3476, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Physical role limitations; Test type: Superiority or Other; p = 0.9045, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Bodily pain; Test type: Superiority or Other; p = 0.8558, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for General health; Test type: Superiority or Other; p = 0.3123, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Vitality; Test type: Superiority or Other; p = 0.3327, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Social functioning; Test type: Superiority or Other; p = 0.8334, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Emotional role limitations; Test type: Superiority or Other; p = 0.7998, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Etanercept BIW vs Etanercept QW; Analysis provided for Mental health; Test type: Superiority or Other; p = 0.7125, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Improvement of Ocular Inflammatory Disease in Patients With Baseline Symptoms
Time Frame: 12 weeks
Population: The population for this assessment was patients who had ocular inflammatory disease at baseline. The number of patients analyzed is zero because no patients had symptoms of ocular inflammatory disease at baseline.
Measure: Number; unit: patients
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in C-reactive Protein (CRP) From Baseline to Week 12.
Description: CRP is a marker of inflammation and measured in mg/l. A higher level is consistent with inflammation.
Time Frame: Baseline and 12 weeks
Population: The analysis population is the intent to treat.
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Etanercept BIW | Etanercept QW
Number analyzed (Participants) | 45 | 44
mg/l | -11.6 (18.42) | -11.7 (21.44)
Statistical Analysis 1: Comparison: Etanercept BIW vs Etanercept QW; Test type: Superiority or Other; p = 0.7404, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Etanercept BIW | Etanercept QW
Serious Adverse Events (participants affected / at risk) | 1 | 2
Other Adverse Events (participants affected / at risk) | 22 | 26
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Etanercept BIW | Etanercept QW
Diarrheic syndrome (Gastrointestinal disorders) | 0/54 | 1/54
Diarrhea (Gastrointestinal disorders) | 1/54 | 0/54
Viral respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0/54 | 1/54
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Etanercept BIW | Etanercept QW
Injection site reaction (General disorders) | 7/54 | 8/54
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5/54 | 8/54
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0/54 | 2/54
Abdominal pain (Gastrointestinal disorders) | 2/54 | 0/54
Diarrhea (Gastrointestinal disorders) | 1/54 | 2/54
Transaminases increased (Investigations) | 4/54 | 4/54
Procedural dizziness (Injury, poisoning and procedural complications) | 1/54 | 2/54
Dizziness (Nervous system disorders) | 2/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.